CLINICAL TRIAL: NCT04851314
Title: Low-flow Anesthesia: Cost-effectiveness of the FLOW-i Anesthesia Machine, a Comparison to Established Anesthesia Delivery Unit
Brief Title: Comparison of Different Ventilator and Vaporizer Technologies to Study Economic and Environmental Implications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Robert Ryan Field, HS/Assistant Clinical Professor; Neuroanesthesiology Clinical Director, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UCIANES11 [HS# 2014-1248]
Record Dates: First submitted 2018-04-30; First posted 2021-04-20 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Anesthetic Gas Consumption and Cost-Effectiveness
Keywords: general anesthesia; anesthesia machines; sevoflurane; low volume ventilator; anesthetic costs; cost-effectiveness; fresh gas flow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ICU certified ventilator (Active Comparator): Participants assigned to receive ventilation with the ICU certified ventilator
  Interventions: Device: ICU certified ventilator
- Non-ICU certified ventilator (Active Comparator): Participants assigned to receive ventilation with the Non-ICU certified ventilator
  Interventions: Device: Non-ICU certified ventilator

INTERVENTIONS:
Device: ICU certified ventilator — Examine anesthetic consumption rates
  Arms: ICU certified ventilator
Device: Non-ICU certified ventilator — Examine anesthetic consumption rates
  Arms: Non-ICU certified ventilator

SUMMARY:
The purpose of this study is to test whether or not the use of a low volume ventilator in an anesthesia machine reduces anesthetic costs significantly as compared to other high volume machines. The study will compare the a low-flow anesthesia machine to a traditional anesthesia machine during routine elective general surgery in patients with ASA ratings of 1-2 under general anesthesia receiving standard care.

DETAILED DESCRIPTION:
The study member will screen for potential subjects using the UCIMC surgical schedule. If a subject is deemed ineligible based on the inclusion and exclusion criteria after reviewing the medical history, his/her record will be discarded. No records will be retained from ineligible subjects. After discussing with the patient's surgeon, study team member will initiate the informed consent process by approaching each eligible subject to explain the study and what it entails. The Lead Researcher will address all questions and concerns from the subject before asking the subject to sign the research consent form.

The GE anesthesia machines currently owned by the operating room will be used to serve as the comparator to the Flow-i machine. The high volume anesthesia machines do not use a low volume system. Subjects will be randomized by recruitment day. On a given recruitment day, all consented subjects will receive anesthesia from one of two groups:

(1) MAQUET FLOW-i device (2) GE anesthetic device

Time points for both groups include:

T0: Time of intubation, when volatile anesthetic are typically first delivered to the patient. We will use 15L/min fresh gas flow, while dictating tidal volumes of 6-8 mL/kg ideal body weight and a PEEP of 6 centimeters of water (cm H2O) in accordance with current best practices.

T1: Time of incision, which typically represents the time of reaching steady state conditions of volatile anesthetic delivery. We will reduce fresh gas flow to 2 L/min in accordance with local practice and weigh the vaporizer at this point, allowing us to measure comparative anesthetic consumption during this wash-in time period (T0-T1).

T2: Time of anesthetic weaning, typically the time when preparing for patient emergence begins by discontinuing the delivery of volatile anesthetics to the patient. The vaporizer will be re- weighed at this point, allowing us to measure comparative anesthetic consumption at steady state maintenance of anesthetic depth (T1-T2) Logically, we will also be able to use T0-T2 in order to understand total comparative anesthetic consumption.

Aside from the randomization to either Group 1 or Group 2, there will be no changes in the surgical or anesthetic procedure, including the medication or treatments given to the subjects as determined by the treating physician. All subjects will receive general anesthesia in accordance to local practice.

For this study, the vaporizer(s) will be weighed on a tared scale before research procedures commence, after induction, and when the gas is shut off during weaning of anesthesia in preparation for extubation to calculate the amount consumed during this time (grams/minute). In addition, the following variables will be recorded:

Subject weight (kg) Tidal Volume (TV) Respiratory Rate (RR) 9 of 24

Positive end-expiratory pressure (PEEP) Fresh Gas Flow Volume % gas End Tidal (%) Time of extubation Time when Aldrete score > 8

This is not a physician-blinded study being that the physical characteristics of the standard delivery units are distinguishable from the MAQUET FLOW-i machine.

All MAC concentrations are standard of care: After the surgical procedure, patient will be assessed for time to reach Aldrete score greater than 8, level of pain and time to extubation. Their medical records will be reviewed to determine need for times and adverse events. Patients will not be contacted for study-related follow-up after they are discharged from recovery.

No photographs or audio/video recording will be collected for this study.

Subject's Privacy:

The study team member will screen for potential subjects using the UCIMC surgical schedule. If a subject is deemed ineligible based on the inclusion and exclusion criteria after reviewing the medical history, his/her record will be discarded. No records will be retained from ineligible subjects.

Study team member will approach each eligible patient to explain the study and what it entails. The study team member will address all questions and concerns from the subjects before asking the patient to sign the research consent form.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Undergo surgery under general anesthesia in UCI Medical Center
* Agree to sign the consent and HIPAA forms
* Subjects who are able to receive sevoflurane

Exclusion Criteria:

* Subjects under the age of 18
* Chronic Obstructive Pulmonary Disease (COPD)
* Body Mass Index (BMI) > 30
* ASA > 2
* Pregnant females
* Procedures less than 2 hours
* Those with known sensitivity to sevoflurane or other halogenated agents; those with known or suspected susceptibility to malignant hyperthermia
* Severe Cardiovascular Disease: Left Ventricular Ejection Fraction (LVEF) < 30%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Field, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avramov MN, Griffin JD, White PF. The effect of fresh gas flow and anesthetic technique on the ability to control acute hemodynamic responses during surgery. Anesth Analg. 1998 Sep;87(3):666-70. doi: 10.1097/00000539-199809000-00033. PMID 9728850
- [Background] Choi SU, Shin HW, Jung HI, Park JY, Yoon SZ, Lee YS, Kim WY, Chang SH. Control of the haemodynamic response to surgical stimuli in semi-closed circuit or closed circuit anaesthesia using a multifunctional anaesthesia system. J Int Med Res. 2010 Sep-Oct;38(5):1637-44. doi: 10.1177/147323001003800508. PMID 21309477

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some enrolled subjects were excluded due to unforeseen circumstances in the clinical workflow e.g. a change in anesthetic preference or canceled surgery. Data from these cases could not provide meaningful results for analysis.
Groups:
- Maquet Flow-i C20: Subjects receiving the Maquet Flow-i C20 anesthetic delivery machine will undergo standardized anesthetic protocol to evaluate anesthetic consumption rates
- GE Aisys CS2: Subjects receiving the GE Aisys CS2 anesthetic delivery machine will undergo standardized anesthetic protocol to evaluate anesthetic consumption rates
Period: Overall Study
Arm/Group | Maquet Flow-i C20 | GE Aisys CS2
Started | 55 | 55
Completed | 52 | 51
Not Completed | 3 | 4
Not completed — Unable to complete research set-up procedures | 0 | 2
Not completed — Change in Anesthesia Plan (patient no longer meets inclusion criteria) | 3 | 2

BASELINE CHARACTERISTICS:
Population: Completed population only
Groups:
- Total: Total of all reporting groups
Arm/Group | Maquet Flow-i C20 | GE Aisys CS2 | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (14) | 44 (13) | 43 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 64
  Male | 17 | 22 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Primary Study Variable: Amount of Gas Vaporized Anesthetic Per Minute Anesthesia
Description: The purpose of this study is to test whether or not the use of a low volume ventilator in an anesthesia machine reduces anesthetic costs significantly as compared to other high volume machines. The study will compare the FLOW-i anesthesia machine to a GE anesthesia machine during routine elective general surgery in patients with ASA ratings of 1-2 under general anesthesia receiving standard care.
Time Frame: Intraoperative (minimum of 2 hours of anesthesia)
Population: Completed patient population for each ventilator type
Measure: Mean (Standard Deviation); unit: grams/minute
Groups:
- Maquet Flow-i C20: Maquet Flow-i C20 (ICU certified ventilator): Examine anesthetic consumption rates
- GE Aisys CS2: GE Aisys CS2 (Non-ICU certified ventilator): Examine anesthetic consumption rates
Arm/Group | Maquet Flow-i C20 | GE Aisys CS2
Number analyzed (Participants) | 52 | 51
grams/minute | 95.48 (49.29) | 119.3 (62.22)

2. Secondary Outcome: Time to Reach Aldrete > 8
Description: Time it took for patient to be safely discharged from the post-anesthesia care unit (PACU).
  The Aldrete Score evaluates recovery after anesthesia and patient readiness to be discharged from PACU. The patient is assessed for consciousness, mobility, breathing, circulation, and color. The evaluation occurs immediately after surgery and then every (1) hour before the patient is deemed ready for discharge.
Time Frame: Up to 24 hours
Population: same as primary outcome measure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Maquet Flow-i C20 | GE Aisys CS2
Number analyzed (Participants) | 52 | 51
minutes | 98.13 (51.83) | 89.18 (52.09)

3. Secondary Outcome: Time to Extubation From Weaning
Description: Time it took to remove patient from mechanical ventilation
Time Frame: Intraoperative (minimum of 2 hours of anesthesia)
Population: same as primary outcome
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Maquet Flow-i C20 | GE Aisys CS2
Number analyzed (Participants) | 52 | 52
minutes | 10.37 (6.321) | 10.78 (6.413)

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 24 hours
Description: As study did not deviate from the standard of care in use of FDA approved devices, any possible adverse event and/or serious adverse event would be the same standard of care.
Arm/Group | Maquet Flow-i C20 | GE Aisys CS2
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 0/52 | 0/51

LIMITATIONS AND CAVEATS:
Some overall limitations include include, but are not limited to: a small overall sample size, fluctuations in the concentration of volatile agent setting or fresh gas flow (due to positioning during surgical preparation), and variations in time precision provider charting of the secondary endpoints (weaning, gas off, time in recovery, recovery criteria completion). Protocol procedures were standardized, however lack of blinding is something the authors could not feasibly account for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT04851314/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT04851314/ICF_001.pdf